CLINICAL TRIAL: NCT06701877
Title: Enhancing Foster Care Relationships Through Attachment-Based Intervention: Protocol of SAFE FAMILY STUDY, a Randomized Controlled Trial of the Circle of Security Parenting® Program in France
Brief Title: Enhancing Foster Care Relationships Through Attachment-Based Intervention: Protocol of SAFE FAMILY STUDY
Acronym: SAFE FAMILIES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shankland Rebecca (Other)
Collaborators: Observatoire National de la Protection de l'Enfance (ONPE) (Unknown); Centre Hospitalier Emile Roux (Other)
Responsible Party: Sponsor-Investigator, Shankland Rebecca, Full Professor of health and developmental psychology, Université Lumière Lyon 2
Organization: Université Lumière Lyon 2 (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SAFE FAMILIES (ULL2/ONPE)
Record Dates: First submitted 2024-11-19; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-10

CONDITIONS: Parenting Sensitivity; Foster Care
Keywords: foster care, Attachment, Circle of Security Parenting intervention, resilience, intervention evaluation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- COSP Intervention Group (Experimental): The intervention group will participate in the COS-P program in addition to TAU. Foster carers will be assigned to groups of 8 to 10 participants and will attend sessions in dedicated training facilities.
  Interventions: Behavioral: Circle of security Parenting (COS-P); Behavioral: Traitement as usual (TAU)
- Waitlist control group (Active Comparator): Waitlist control groupe will continue to receive Treatment as Usual (TAU), which consists of Psycho-Educational Support (PSE) provided by Child Protection Services. PSE typically involves home visits, educational and psychological support for foster carers and/or children in placement, and efforts to support and monitor contact between children and their birth families. The control group will be placed on a waiting list to receive the COS-P program as part of continuing education at a later date.
  Interventions: Behavioral: Traitement as usual (TAU)

INTERVENTIONS:
Behavioral: Circle of security Parenting (COS-P) — The Circle of Security Parenting® (COS-P) program is an attachment-based intervention designed to enhance caregiver sensitivity, parental reflective functioning, and the quality of the child's attachment to their caregiver. This manualized intervention, with both educational and therapeutic components, empowers caregivers to better understand and respond to their child's needs, fostering secure attachment (22).
  Arms: COSP Intervention Group
Behavioral: Traitement as usual (TAU) — TAU typically involves home visits, educational and psychological support for foster carers and/or children in placement, and efforts to support and monitor contact between children and their birth families.

SUMMARY:
Background: Children in out-of-home care constitute a vulnerable population often experiencing mental health challenges related to early adversity and placement disruptions. The Circle of Security Parenting® (COS-P) program is an attachment-based intervention designed to enhance carer sensitivity and reflective functioning, ultimately improving the quality of carer-child relationships.

Methods This study protocol follows a mixed-methods randomized controlled trial evaluating the effectiveness of the COS-P program for foster carers in France. A total of 70 foster carers will be randomly assigned to either the intervention group (receiving COS-P in addition to Treatment as Usual) or the waitlist control group (receiving Treatment as Usual only). Quantitative measures, including the Caregiving Composite Questionnaire, Parenting Stress Index, and the Marschak Interaction Method, will be administered at baseline and at follow-up). Qualitative data will be collected through focus groups with foster carers and COS-P facilitators, and through self-confrontation interviews with a subset of foster carers.

Discussion: This study is the first to evaluate COS-P for foster carers in France. Findings will provide valuable insights into the program's effectiveness in improving carer-child relationships and foster carer well-being, ultimately contributing to better outcomes for children in out-of-home care. The study will also explore potential moderators of treatment outcome and shed light on the subjective experiences of participants.

ELIGIBILITY:
Inclusion Criteria:

Foster carers:

1. Signed informed consent form.
2. Commitment to attend all eight sessions of the COS-P program.
3. Employed by CPS Haute-Loire or by one of the two participating private agencies.

Foster children:

1. Placed with a foster carer participating in the study.
2. Aged from 1 to 6 years.
3. In permanent placement (5 or more days per week with the foster carer).
4. Consent obtained from all individuals holding parental responsibility.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Caregiving composite questionnaire (CCQ) | at baseline and at 3 month f/u
  The CCQ is a 43-item self-report measure specifically designed to assess parent capacities targeted by the COS-P program, namely: parental mentalizing, parenting self-efficacy, and parent perceptions of the child. It combines six subscales and one single item drawn from previously validated measures, retaining the original response formats and scoring procedures for each subscale. The CCQ has demonstrated good reliability and validity in a pilot sample of parents and is being used in the current study to assess the impact of COS-P on these key parenting capacities.
Parent Development Interview-Revised | At baseline and at 3-month f/u
  This semi-structured interview consists of 31 questions, administered in approximately one hour, covering four domains: (a) perception of the child, (b) perception of the relationship, (c) parental affective experience, and (d) separation experiences.

SECONDARY OUTCOMES:
Parenting Stress Index - IV - Short Form (PSI) | At baseline and 3-month f/u
  This 36-item questionnaire includes three subscales: Parental Distress (PD), Parent-Child Dysfunctional Interaction (P-CDI), and Difficult Child (DC). The 12 items of the P-CDI subscale will be used to assess foster carers' perceptions of their relationship with the child in their care, using a 5-point Likert scale.
Marschak Interaction Method (MIM) | At baseline and 3-month f/u
  This structured assessment tool is based on attachment and mentalization theories and involves a series of age-appropriate tasks completed by the foster carer and child together. The MIM assesses four dimensions of interaction: Structure, Engagement, Nurture, and Challenge. Interaction recordings will be coded using the Dyadic Emotional Interaction Style (D-EIS), developed in Finland and used internationally.

CONTACTS AND LOCATIONS:
Locations (1):
- DEPARTEMENT de la Haute-Loire, Le Puy-en-Velay, France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maxwell AM, McMahon C, Huber A, Hawkins E, Reay RE. Addressing the Evidence Gap: Protocol for an Effectiveness Study of Circle of Security Parenting, an Attachment-Based Intervention. Front Glob Womens Health. 2020 Oct 22;1:575752. doi: 10.3389/fgwh.2020.575752. eCollection 2020. PMID 34816157
- [Background] Helle J, Vollestad J, Schanche E, Hjelen Stige S. From seeing difficult behaviour to recognizing legitimate needs - A qualitative study of mothers' experiences of participating in a Circle of Security Parenting program in a public mental health setting. Psychother Res. 2023 Apr;33(4):482-493. doi: 10.1080/10503307.2022.2132888. Epub 2022 Oct 31. PMID 36314235
- [Background] Engler AD, Sarpong KO, Van Horne BS, Greeley CS, Keefe RJ. A Systematic Review of Mental Health Disorders of Children in Foster Care. Trauma Violence Abuse. 2022 Jan;23(1):255-264. doi: 10.1177/1524838020941197. Epub 2020 Jul 20. PMID 32686611
- [Derived] Pereira M, Sedes L, Gadea E, Shankland R. Enhancing foster care relationships through attachment-based intervention: the safe families study protocol, a randomized controlled trial of the circle of security parenting program(R). BMC Psychol. 2025 Feb 8;13(1):107. doi: 10.1186/s40359-025-02424-6. PMID 39923102